CLINICAL TRIAL: NCT07256015
Title: "DEMOS" - Deucravacitinib for Patients With Moderate/Severe Psoriasis: A Real-Life Experience in Italy
Brief Title: Deucravacitinib for Patients With Moderate/Severe Psoriasis: A Real-Life Experience in Italy
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1228
Record Dates: First submitted 2025-08-28; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
Keywords: Moderate/Severe Psoriasis
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular | interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with moderate/severe psoriasis receiving deucravacitinib
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — According to the product label

SUMMARY:
The purpose of this study is to characterize the real-life experience of patients with moderate/severe psoriasis receiving deucravacitinib treatment, in terms of efficacy, safety, and health-related quality of life (HRQoL) in Italy

ELIGIBILITY:
Inclusion Criteria:

* Participants have initiated treatment with deucravacitinib monotherapy 4 to 8 weeks earlier according to clinical practice and to reimbursement criteria determined by National Drug Agency in Italy (AIFA)
* Patients have moderate to severe plaque psoriasis
* Patients have signed informed consent form (ICF)

Exclusion Criteria:

* Simultaneous participation in any interventional study for their moderate-to-severe psoriasis
* Inability to participate to the study for the following reasons: patients unable to understand the aim of the study, patients unable to understand and sign the ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults diagnosed moderate/severe psoriasis who have already started treatment with deucravacitinib according to clinical practice and to reimbursement criteria determined by the National Drug Agency (AIFA) in Italy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-07-05 (Estimated); Study Completion 2027-08-05 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants still receiving deucravacitinib treatment | Week 24 and 52
Absolute Psoriasis Area and Severity Index (PASI) | Baseline and Weeks 16, 24 and 52

SECONDARY OUTCOMES:
Participant age in years | Baseline
Participant sex | Baseline
Participant height in cm | Baseline
Participant body mass index in kg/m2 | Baseline
Participant previous pathologies | Baseline
Participan previous surgical procedures | Baseline
Date of psoriasis diagnosis | Baseline
Number of participants with physical examination according to body systems | Baseline
Participant treatment history | Baseline
  Treatment history to describe participants previous treatment(s) received for psoriasis and participants previous treatment(s) received not related to psoriasis
Participant comorbidities | Baseline
Quality of life as assessed by the Dermatology Life Quality Index (DLQI) questionnaire | Baseline and Weeks 16, 24 and 52
Change in symptoms as assessed by the Itch Numerical Rating Scale (Itch-NRS) score | Baseline and Weeks 16, 24 and 52
Body Surface Area (BSA) | Baseline and Weeks 16, 24 and 52
Static Physician's Global Assessment (sPGA) score | Baseline and Weeks 16, 24 and 52
Scalp Specific Physician Global Assessment (ssPGA) score | Baseline and Weeks 16, 24 and 52
Scalp Specific Physician Global Assessment (ssPGA) score 0/1 | Baseline and Weeks 16, 24 and 52
Absolute Psoriasis Area and Severity Index (PASI) 75 and 90 | Baseline and Weeks 16, 24 and 52
Concomitant psoriasis therapies received | Baseline and Weeks 16, 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts